CLINICAL TRIAL: NCT00144898
Title: A Randomized, Phase III Clinical Trial GF-GS 01 to Compare Conventional Axillary Dissection Versus Sentinel Node Resection (GS) in Clinically Node-negative Operable Breast Cancer Unifocal N0 Patients
Brief Title: GF-GS 01: Comparing Conventional Axillary Dissection Versus Sentinel Node Resection in Clinically Node-negative Operable Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.312
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; sentinel node resection; survival; Breast cancer unifocal N0
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sentinel Node Resection (Experimental): Sentinel Node Resection
  Interventions: Procedure: Sentinel Node Resection
- Conventional Axillary Dissection (Other): Conventional Axillary Dissection
  Interventions: Procedure: Conventional Axillary Dissection

INTERVENTIONS:
Procedure: Sentinel Node Resection — Sentinel Node Resection
  Arms: Sentinel Node Resection
Procedure: Conventional Axillary Dissection — Conventional Axillary Dissection
  Arms: Conventional Axillary Dissection

SUMMARY:
Sentinel node resection appears as a promising advancement in the surgical treatment of breast cancer.

The GF-GS 01 study, sponsored by a National Hospital Research Program, compares this new surgical method with a classical method in patients having a negative sentinel node.

The duration of the follow-up is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years with clinically node-negative operable unifocal N0 breast cancer (clinical tumour size < 30 mm).
* Written consent is obtained from all patients before randomization.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1627 (Actual)
Dates: Start 2003-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Survival without recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles HOUVENAEGHEL, MD, Principal Investigator — Institut Paoli Calmette
Locations (1):
- Alain LEIZOROVICZ, Lyon, France

REFERENCES:
- [Result] Roy P, Leizorovicz A, Villet R, Mercier C, Bobin JY. Systematic versus sentinel-lymph-node-driven axillary-lymph-node dissection in clinically node-negative patients with operable breast cancer. Results of the GF-GS01 randomized trial. Breast Cancer Res Treat. 2018 Jul;170(2):303-312. doi: 10.1007/s10549-018-4733-y. Epub 2018 Mar 10. PMID 29526019